CLINICAL TRIAL: NCT01512368
Title: Changes in Serum Fibroblast Growth Factor 21 (FGF21) Levels After a Cardiorespiratory Exercise Program
Brief Title: Changes in Serum Fibroblast Growth Factor 21 (FGF21) Levels Correlated With Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Daniel Cuevas-Ramos, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: REF173; 48024 (Other Grant/Funding Number: Consejo Nacional de Ciencia y Tecnología (CONACYT)/216324)
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Sedentary Lifestyle
Keywords: Fibroblast growth factor 21 (FGF21); Exercise; Metabolic equivalents (METs); Lipolysis; Glucose; Free fatty acids (FFAs); Epinephrine
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supervised exercising (Experimental): A treadmill exercise test (following the Bruce's protocol) was done five times per week (from Monday to Friday) for two weeks to participants.
  Interventions: Other: Supervised Exercising

INTERVENTIONS:
Other: Supervised Exercising — A treadmill exercise test (following the Bruce's protocol) was done five times per week (from Monday to Friday) for two weeks.
  Other Names: Bruce's protocol

SUMMARY:
We evaluated the effect of two weeks of intensive supervised physical activity in serum fibroblast growth factor 21 (FGF21) levels.

DETAILED DESCRIPTION:
Comparative and longitudinal study. Anthropometric and biochemical evaluation were done before, 1hr and 4hr after a bout of exercise and repeated after two weeks of daily supervised exercise. We studied sedentary young healthy women. A treadmill exercise test (following the Bruce's protocol) was done five times per week (from Monday to Friday) for two weeks. The Department of Endocrinology and Metabolism at the INCMNSZ performed all biochemical laboratory measurements using standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Aged 18 to 35 years old,
* Body mass index (BMI) <30 kg/m2
* Without contraindication for exercising

Exclusion Criteria:

* Metabolic syndrome
* Diabetes
* Dyslipidemia
* Hypertension
* Asthma
* Thyroid disease
* Treated with fibrates, beta agonists or blockers
* History or current arrhythmias, murmurs, cardiomegaly, or treatment for cardiovascular diseases -
* Contraindications for exercise testing were also considered as exclusion criteria (see references)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cuevas-Ramos, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Paloma Almeda-Valdes, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Carlos A Aguilar-Salinas, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- INCMNSZ, Mexico City, Tlalpan, Mexico

REFERENCES:
- [Background] Cuevas-Ramos D, Almeda-Valdes P, Gomez-Perez FJ, Meza-Arana CE, Cruz-Bautista I, Arellano-Campos O, Navarrete-Lopez M, Aguilar-Salinas CA. Daily physical activity, fasting glucose, uric acid, and body mass index are independent factors associated with serum fibroblast growth factor 21 levels. Eur J Endocrinol. 2010 Sep;163(3):469-77. doi: 10.1530/EJE-10-0454. Epub 2010 Jun 21. PMID 20566587
- [Background] Hill J, Timmis A. Exercise tolerance testing. BMJ. 2002 May 4;324(7345):1084-7. doi: 10.1136/bmj.324.7345.1084. No abstract available. PMID 11991917
- [Derived] Cuevas-Ramos D, Almeda-Valdes P, Meza-Arana CE, Brito-Cordova G, Gomez-Perez FJ, Mehta R, Oseguera-Moguel J, Aguilar-Salinas CA. Exercise increases serum fibroblast growth factor 21 (FGF21) levels. PLoS One. 2012;7(5):e38022. doi: 10.1371/journal.pone.0038022. Epub 2012 May 31. PMID 22701542
- See also: INCMNSZ — http://www.innsz.mx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2010 to August 2011 a total of 60 sedentary young women without contraindication for exercising were included. Study was carried out at Department of Endocrinology, Cardiology and Internal Medicine of the INCMNSZ.
Pre-assignment Details: In the initial visit, patients were instructed to keep unaltered their diet, lifestyle and physical activity. Basal daily physical activity was evaluated with a questionnaire. All participants were assigned to the intervention group. All subjects underwent basal and final physical and biochemical evaluation.
Period: Overall Study
Arm/Group | Supervised Exercising
Started | 63
Completed | 60
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.0 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 63

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Fibroblast Growth Factor 21 (FGF21) Acutely and at Two Weeks
Description: Serum measurement of FGF21 using human ELISA kit was done at baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise.
Time Frame: Baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Population: The sample size was calculated using the formula for means for two-tailed comparisons. According to our previous report, we expected a minimal change of 80 ng/l of FGF21 after two weeks of physical activity. Using a SD of 160 ng/l with an alfa of 0.05 and a study power of 80%, a total of 60 subjects were calculated. All participants were analyzed.
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 60
ng/L
  Baseline | 276.8 [142.8 to 568.6]
  Final (after 2 weeks) | 460.8 [298.2 to 742.1]
Statistical Analysis 1: Comparison: Supervised Exercising; FGF21 was log transformed to approximate normality before analyses. Null hypothesis was Ho = Y1 (FGF21 level at baseline) = Y2 (FGF21 level after two weeks of exercising). Power calculation was 80% with 60 participants evaluated (one group). To evaluate the effect of exercise on clinical and biochemical parameters, we used the difference between final - basal levels ("delta"); Test type: Superiority or Other; p < 0.001, Regression, Linear — All reported p values are based on two-sided tests considering ≤0.05 as significant; Adjusted for age, time of exercise, creatinine, waist to hip ratio, fat percentage, body mass index, mean rest heart rate, blood pressure; Slope = 0.089, 95% CI 2-sided [0.034 to 0.144], Standard Error of Mean 0.063 — Metabolic equivalents (METs) consumed were independently associated with the log of delta (final-basal) FGF21 levels

2. Secondary Outcome: Change From Baseline Free Fatty Acids (FFAs) Acutely and at Two Weeks
Description: Serum measurement of free fatty acids (FFAs) was done at baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise.
Time Frame: Baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Population: The sample size was calculated using the formula for means for two-tailed comparisons. According to our previous report, we expected a minimal change of 80 ng/l of FGF21 after two weeks of physical activity. Using a SD of 160 ng/l with an alfa of 0.05 and a study power of 80%, a total of 60 subjects were calculated.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 60
mg/dL
  Baseline | 0.36 [0.24 to 0.44]
  Final (after 2 weeks) | 0.54 [0.43 to 0.66]

3. Secondary Outcome: Change From Baseline Epinephrine Acutely and at Two Weeks
Description: Serum measurement of epinephrine was done at baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise.
Time Frame: Baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Population: The sample size was calculated using the formula for means for two-tailed comparisons. According to our previous report (5), we expected a minimal change of 80 ng/l of FGF21 after two weeks of physical activity. Using a SD of 160 ng/l with an alfa of 0.05 and a study power of 80%, a total of 60 subjects were calculated.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 60
pg/mL
  Baseline | 9.2 [5.9 to 12.1]
  Final (at 2 weeks) | 15.5 [11.3 to 18.8]

4. Secondary Outcome: Change From Baseline Leptin Acutely and at Two Weeks
Description: Serum measurement of leptin was done at baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Time Frame: Baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 60
ng/mL
  Baseline | 13.1 [8.7 to 21.1]
  Final (at 2 weeks) | 12.4 [10.0 to 16.2]

5. Secondary Outcome: Change From Baseline Total Adiponectin Acutely and at Two Weeks
Description: Serum measurement of total adiponectin was done at baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Time Frame: Baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 60
ng/mL
  Baseline | 10.1 [8.0 to 13.4]
  Final (at 2 weeks) | 10.5 [8.0 to 13.2]

6. Secondary Outcome: Change From Baseline Fasting Glucose Acutely and at Two Weeks
Description: Serum measurement of glucose was done at baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Time Frame: Baseline, 1hr and 4 hr after a bout of exercise, and repeated after two weeks of daily supervised exercise
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Supervised Exercising
Number analyzed (Participants) | 60
mg/dL
  Baseline Glucose | 86.0 (7.1)
  Final Glucose (at 2 weeks) | 86.3 (6.4)

ADVERSE EVENTS:
Time Frame: Adverse events were supervised throughout every treadmill test.
Description: Continuous electrocardiographic monitoring were registered in every treadmill test.
Arm/Group | Supervised Exercising
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

LIMITATIONS AND CAVEATS:
We cannot fully control other potential sources of physical activity. The results may not be applicable to men. We did not register the caloric consumption during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No